CLINICAL TRIAL: NCT02923297
Title: GALIG Gene Expression in Parkinson's Disease
Acronym: GALIGPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: National Scientific Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2014-05
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
Keywords: parkinson; alpha-synuclein; GALIG; quantitative PCR (polymerase chain reaction)
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parkinson's disease patients (Other): blood sampling
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — blood sampling for determine and compare the expression patterns of GALIG gene

SUMMARY:
Parkinson's disease (PD) is the most frequent neurodegenerative disorder after Alzheimer's disease. It is characterized by motor symptoms (rigidity, tremor, slowness of movements), and non-motor symptoms (neuropsychological, psychiatric, pain ...). Neuronal death initiates in the brainstem and extends progressively through the entire cortex. The processes leading to cell death are poorly understood. Pathological cells exhibit abnormal deposits, called Lewy bodies, which contain numerous proteins. A major constituent of these protein deposits is alpha-synuclein. It has recently been demonstrated, in the Laboratory of Molecular Biophysics of the CNRS (Scientific Research National Center) in Orleans, that α-synuclein interacts with Cytogaligin, a protein produced by the proapoptotic GALIG gene. Cytogaligin could thus be a factor regulating α-synuclein activity or aggregation. It is postulated that the level of expression of the GALIG gene is different in Parkinson's disease patients compared with control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease according to the criteria of the UKPDBB (UK Parkinson's disease brain bank).

Exclusion Criteria:

* Insane patient arriving without a third party.
* Patient with Parkinson's disease arising from another etiology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
RNA (ribonucleic acid) assay of GALIG gene | Day 0
  Only one assessment in the study
RNA (ribonucleic acid) assay of SNCA genes | Day 0
  Only one assessment in the study

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, Ph, Principal Investigator — CHR d'ORLEANS
Locations (1):
- CHR d'ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alieva AKh, Filatova EV, Karabanov AV, Illarioshkin SN, Slominsky PA, Shadrina MI. Potential Biomarkers of the Earliest Clinical Stages of Parkinson's Disease. Parkinsons Dis. 2015;2015:294396. doi: 10.1155/2015/294396. Epub 2015 Sep 21. PMID 26483988
- [Background] Pinho R, Guedes LC, Soreq L, Lobo PP, Mestre T, Coelho M, Rosa MM, Goncalves N, Wales P, Mendes T, Gerhardt E, Fahlbusch C, Bonifati V, Bonin M, Miltenberger-Miltenyi G, Borovecki F, Soreq H, Ferreira JJ, F Outeiro T. Gene Expression Differences in Peripheral Blood of Parkinson's Disease Patients with Distinct Progression Profiles. PLoS One. 2016 Jun 20;11(6):e0157852. doi: 10.1371/journal.pone.0157852. eCollection 2016. PMID 27322389
- [Background] Scherzer CR, Eklund AC, Morse LJ, Liao Z, Locascio JJ, Fefer D, Schwarzschild MA, Schlossmacher MG, Hauser MA, Vance JM, Sudarsky LR, Standaert DG, Growdon JH, Jensen RV, Gullans SR. Molecular markers of early Parkinson's disease based on gene expression in blood. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):955-60. doi: 10.1073/pnas.0610204104. Epub 2007 Jan 10. PMID 17215369